CLINICAL TRIAL: NCT03213561
Title: Stable and Independent Non-invasive Communication Brain-computer Interfaces Based on Error-adaptive Decoding Algorithms
Brief Title: Stable and Independent Communication Brain-computer Interfaces
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have not succeeded in developing an approach that uses hdEEG to control a communication interface at an accuracy needed to complete the protocol.
Sponsor: Tomislav Milekovic (Other)
Collaborators: University of Geneva, Switzerland (Other); Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other); Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Sponsor-Investigator, Tomislav Milekovic, Principal Investigator, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-00639
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Tetraplegia; Locked-in Syndrome
MeSH Terms: conditions — Quadriplegia; Locked-In Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stable and Independent Communication Brain-computer Interfaces (Experimental): Each arm will receive the same intervention.
  Interventions: Device: Stable and Independent Brain-computer Interfaces for Communication

INTERVENTIONS:
Device: Stable and Independent Brain-computer Interfaces for Communication — The participants will perform an MRI head scan, which the investigators will use to construct 3D head models of participants. The investigators will use these modele to reconstruct the activity of brain sources from EEG signals. The participants will then take part in a series of EEG recording sessions. During the initial "calibration" sessions, the participants will react with real or attempted movements to visual cues. The investigators will use the EEG signals from these sessions to calibrate the text-entry interface used in the validation sessions that follow. During the validation sessions, the participants will control the text-entry interface to write messages using their EEG signals.

SUMMARY:
People with locked-in syndrome cannot move their limbs or talk because of a motor impairment, but remain conscious and intellectually awake. Restoring the ability to communicate to people with locked-in syndrome will have a positive effect on their quality of life, will enable them to reintegrate into society and increase their capacity to lead productive and fulfilling lives. This study sims to develop a new assisted communication device based on a brain-computer interface, a system that allows the user to control a computer with his brain activity. The investigators will develop this brain-computer system for long-term stability and independent use by using adaptive decoders. The investigators will test the long-term stability and independence of this system with healthy volunteers, people with tetraplegia and people with locked-in syndrome over time periods of several months.

ELIGIBILITY:
Inclusion criteria for healthy persons:

* Older than 18
* Fluent in French, English, German or Italian
* Good visual acuity

Inclusion criteria for people with tetraplegia:

* Older than 18
* Fluent in French, English, German or Italian
* Good visual acuity
* Diagnosed with spinal cord injury, brainstem stroke, spinal stroke, muscular dystrophy or other non-degenerative motor neuron disorders
* Limited or no ability to use both hands - less than grade 4 muscle strength in elbow extension and wrist extension and less than grade 2 strength in finger flexor and abduction on both sides

Inclusion criteria for people with locked-in syndrome:

* Were fluent in French, English, German or Italian before losing the ability to speak
* Enough visual capability to see large letters from a distance of around 50cm according to caretaker's or guardian's opinion

Exclusion criteria for healthy persons:

* Smokers
* Substance or alcohol abuse
* Neurological or psychiatric illness
* History of cranio-facial surgery
* Metallic implants that would prohibit the subject from having a MRI scan
* Medications that may retard motor coordination and cognitive ability (such as sedatives)
* Seizure disorders
* Treated with anti-epileptic medications

Exclusion criteria for people with tetraplegia and locked-in syndrome:

* Disabling neurological illness other than tetraplegia or locked-in syndrome
* Disabling psychiatric illness
* History of cranio-facial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Brain-computer interface stability | 3 years
  The investigators will measure the text-entry rate achieved using the brain-computer interface in each session by the number of correct characters per minute (CCPM). At the end of the study, the investigators will calculate the average brain-computer interface performance, and the correlation between the performance and the duration of brain-computer interface use (performance-use correlation). Brain-computer interface stability will be established if the performance-use correlation is greater than -0.5 CCPM/year. Primary objective of the study will be met if the brain-computer interface performance is stable for 75% of participants or more in each of three study populations, and if the average brain-computer interface performance for participants that show stable performance is greater than 5 CCPM.

SECONDARY OUTCOMES:
Brain-computer interface performance comparison | 3 years
  At the end of the study, the investigators will compare the brain-computer interface performance and the performance-use correlation between the three study populations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Campus Biotech, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No